CLINICAL TRIAL: NCT02270021
Title: Randomized Trial to Increase Adherence to Cervical Cancer Screening Guidelines for Young Women
Brief Title: Decreasing Over Screening and Treatment of Cervical Precancers in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Latinas Contra Cancer (Unknown); National Cervical Cancer Coalition (Unknown); California Department of Health Services (Other); American College of Obstetricians and Gynecologists (Other); American Society for Colposcopy and Cervical Pathology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 13-12257; CD-1304-6551 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Cervical Cancer
Keywords: Pap smear; Screening; Women; Human papillomavirus; Cervical precancer; Guideline adherence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: clinic sites were randomized not subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Provider Mobile Application (ProvAPP) (Experimental): Mobile phone application for providers.
  Interventions: Other: Provider Mobile Application (ProvAPP)
- ProvAPP + Patient Educational Tool (Tab) (Experimental): Patient educational tool; plus the Mobile phone application for providers.
  Interventions: Other: ProvAPP + Patient Educational Tool (Tab)
- ProvAPP Control Group (No Intervention): Clinics in this group are those NOT randomized - receiving no intervention. These clinics will be chosen at random for comparison using Family PACT claims data.
- ProvAPP+Tab Control Group (No Intervention): Clinics in this group are those NOT randomized - receiving no intervention. These clinics will be chosen at random for comparison using Family PACT claims data.

INTERVENTIONS:
Other: Provider Mobile Application (ProvAPP) — Mobile phone application to maneuver clinicians through the cervical cancer screening and treatment guidelines based on patient age and condition.
  Arms: Provider Mobile Application (ProvAPP)
Other: ProvAPP + Patient Educational Tool (Tab) — Patient Educational Tool (Tab): A patient educational tool (mobile tablet) will educate women on cervical cancer screening and treatment. Patients' self-assessment using a tablet at the time of clinic check-in will help them to understand current guidelines and their choices for treatment if they have abnormal cytology. It will allow them to assess the risks and benefits of screening intervals and of treatment choices.
  ProvAPP: Mobile phone application to maneuver clinicians through the cervical cancer screening and treatment guidelines based on patient age and condition.
  Arms: ProvAPP + Patient Educational Tool (Tab)

SUMMARY:
The goal of this study is to prevent over screening and over treatment of young women for cervical precancers, which can result in psychological distress and has been associated with future risk of premature deliveries. Current national guidelines recommend that routine screening be performed at less-frequent intervals and that excisional cervical therapies are discouraged in young women. The objectives of this study are to examine physician- and patient-based interventions designed to decrease over screening and over treatment by increasing adherence to US guidelines for women under 30 years.

DETAILED DESCRIPTION:
In this study, we compare two different intervention arms that are designed to prevent over screening and over treatment by increasing adherence to the new US cervical cancer screening guidelines and the American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines for the management of abnormal cervical cancer screening tests and cancer precursors. Specifically, the interventions will focus on the newly recommended cervical cancer screening intervals and decreasing the number of colposcopy procedures and cervical procedures for abnormal cytology.

This is a cluster randomized trial with individual clinics serving as the clusters. Clinics from the California Family PACT provider network who serve at least 200 female clients per year under 30 years of age will be randomized to one of two arms: 1) ASCCP mobile application (ProvAPP)-based intervention for providers, or 2) ProvAPP + Patient education Tool (Tab) intervention. These groups will be compared to a control comparison group of 28 clinics chosen using propensity score matching based on clinic characteristics such as county and private versus public from the Family PACT claims data. The ProvAPP intervention is for clinicians' mobile phones and will help them maneuver through current guidelines based on patient age and condition. An existing application from the ASCCP will be updated to include screening guidelines and to be more user-friendly. The patient-based Tab intervention will be a patient education tool accessible via URL on a tablet device at the time of check-in to assist in asking questions and evaluating treatment options. The tool will be developed with input from women age 21-29 as well as other stakeholders including Latinas Contra Cancer and the National Cervical Cancer Coalition. It is hypothesized that the ProvAPP+Tab approach will be most successful; all interventions will be more successful than no intervention.

Family PACT serves predominantly uninsured women and 40% of clients are Latina. We plan to enroll 7 sites (ProvAPP) and 7 sites (ProvAPP+Tab) into the other intervention arm with an average of 2,800 women to 3,500 women aged 21-29 years per arm (14 sites) with a similar number of sites and women randomly chosen for the comparison arm (28 sites) resulting in a total of 39 sites and 8,400-10,500 women. We will use Family PACT claims data to examine, by age, the number of and average interval between cytology specimens, colposcopy examinations, and the number of excisional procedures.

ELIGIBILITY:
Inclusion Criteria - Patients:

* English or Spanish speaking
* Women
* Age 21-29 years
* History of one or more of the following: abnormal Pap smear, normal Pap smear, no Pap smear, cervical cancer

Exclusion Criteria - Patients:

* Language other than English or Spanish
* Male
* Younger than 21 or older than 29

Inclusion Criteria - Clinics:

* Family PACT provider
* Not a Planned Parenthood affiliate
* Located in one of ten identified Southern California study counties
* Sends cytology/histology specimens to Quest Diagnostics West Hills
* Clinical care visits occurred to at least 200 women age 21-29 years in fiscal year 2011/2012
* Has a calculated average cytology interval of less than 30 months (based on last three years)

Exclusion Criteria - Clinics:

* Not a Family PACT provider
* Planned Parenthood affiliate
* Not located in one of ten identified Southern California study counties
* Sends cytology/histology specimens to a lab other than Quest Diagnostics West Hills
* Clinical care visit occurred to less than 200 women age 21-29
* Has a calculated average cytology interval of more than 30 months

Ages: 21 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of Cervical Cancer Screening | Change from baseline screening rate (3 months prior to intervention) to 15-18 months after start of intervention
  Rate of women 21-29 years who received cervical cytology tests.

SECONDARY OUTCOMES:
Rate of Colposcopy | Change from baseline colposcopy rate (3 months prior to intervention) to 15-18 months after start of intervention
  Rate of women 21-29 years who receive colposcopy for cervical cancer screening over the total number of women 21-29 years.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Barbara Moscicki, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Derived] Moscicki AB, Chang C, Vangala S, Zhou X, Elashoff DA, Dehlendorf C, Sawaya GF, Kuppermann M, Duron Y, Wyand FL, Navarro SK, Thiel de Bocanegra H. Effect of 2 Interventions on Cervical Cancer Screening Guideline Adherence. Am J Prev Med. 2021 May;60(5):666-673. doi: 10.1016/j.amepre.2020.11.015. Epub 2021 Feb 23. PMID 33632649

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT02270021/Prot_SAP_000.pdf